CLINICAL TRIAL: NCT00581360
Title: Phase II Trial of Doxorubicin and Bortezomib in Patients With Incurable Head and Neck Adenoid Cystic Carcinoma
Brief Title: Phase II Trial of Doxorubicin and Bortezomib in Patients With Incurable Adenoid Cystic Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-124
Record Dates: First submitted 2007-12-19; First posted 2007-12-27 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Adenoid Cystic Carcinoma
Keywords: Adenoid cystic carcinoma; bortezomib; doxorubicin
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — Doxorubicin; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib + Doxorubicin (Other): Patients with incurable adenoid cystic carcinoma of the head and neck who receive doxorubicin and bortezomib
  Interventions: Drug: doxorubicin and bortezomib

INTERVENTIONS:
Drug: doxorubicin and bortezomib — Patients will be treated with bortezomib 1.3 mg/m2, intravenously on days 1, 4, 8 and 11, and doxorubicin 20 mg/m2, intravenously on days 1 and 8, every 21 days. Zinecard will be added at the 8th cycle and all subsequent cycles with doxorubicin. After the completion of 14 cycles, if there is no progression, bortezomib once a week at a dose of 1.6 mg/m2 on days 1,8,15, every 28 days, will be administered alone. Treatment will continue unless disease progression or intolerable toxicity emerges.
  Other Names: Velcade

SUMMARY:
This is a Phase II trial non-randomized study to evaluate the objective response rate and stable disease rate (primary endpoints), progression-free survival, overall survival and toxicities with the combination of doxorubicin and bortezomib in patients with incurable head and neck adenoid cystic carcinoma. Also, we plan to collect tumor tissue from previous diagnostic procedures and baseline blood specimens for future correlative studies.

DETAILED DESCRIPTION:
Patients will be treated with bortezomib 1.3 mg/m2, intravenously on days 1, 4, 8 and 11, and doxorubicin 20 mg/m2, intravenously on days 1 and 8, every 21 days. Zinecard will be added at the 8th cycle and all subsequent cycles with doxorubicin. After the completion of 14 cycles, if there is no progression, bortezomib once a week at a dose of 1.6 mg/m2 on days 1,8,15, every 28 days, will be administered alone. Treatment will continue unless disease progression or intolerable toxicity emerges (see section 5 for detailed treatment plan and dose modifications).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have locally advanced, recurrent, or metastatic adenoid cystic carcinoma of the head and neck which is considered incurable by known therapies, as judged by the investigator.
* Patients should have cytologically or histologically confirmed adenoid cystic carcinoma of the head and neck.
* Patients must have unidimensionally measurable disease (RECIST criteria). If the only site of measurable disease is a previously irradiated area, the patient must have documented progression of disease in this area.
* All available prior computed tomography (CT) or magnetic resonance imaging (MRI) scans should be reviewed and noted, and measurements showing progression of disease should be documented whenever possible. However, documentation of disease progression is not mandatory for enrollment.
* Patients must have multigated acquisition scan (MUGA) scan showing left ventricular ejection function (LVEF) at or above the institutional lower limits of normal.
* Patients must have ECOG performance status 0-2.
* Patients should have recovered from prior surgery or radiation therapy. A minimum time period of 3 weeks should elapse between the completion of extensive radiation therapy for recurrent/metastatic disease and enrollment in the study.
* Patients must have normal organ and marrow function (as defined below) measured within one week prior to registration:
* Absolute neutrophil count >1,500/mm3.
* Platelets greater than or equal to 100,000/mm3.
* Total bilirubin within normal institutional limits.
* Transaminases (AST and ALT) <3 X ULN.
* Creatinine within normal institutional limits or creatinine clearance (CrCl) greater than or equal to 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal. CrCl will be calculated using the Cockcroft-Gault formula:
* Calculated Creatinine Clearance = (140-age) X actual body wt.(kg) 72 X serum creatinine. Multiply this number by 0.85 if the patient is female.
* Myocardial infarction within 6 months prior to enrollment, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant. Patients must not have history of congestive heart failure of any grade according to Heart Association (NYHA) (see Appendix 2).
* Age > 18 years and capacity to give informed consent.
* All patients must have given signed, informed consent prior to registration to the study.

Exclusion Criteria:

* No prior chemotherapy for recurrent / metastatic adenoid cystic carcinoma. Up to 1 prior biologic/targeted therapy regimen is allowed. Also, chemotherapy as part of initial potentially curative therapy (i.e. concurrent chemoradiotherapy) is allowed, if it was completed >6 months earlier.
* Patients must not have any prior anthracyclines (doxorubicin, epirubicin, daunorubicin, idarubicin) or mitoxantrone, or bortezomib.
* No history of prior malignancy, with the exception of curatively treated squamous cell or basal carcinoma of the skin or in situ cervical cancer, unless there is a 3-year disease-free interval.
* Patients must not have history of allergic reactions attributed to compounds of similar chemical or biologic composition to bortezomib, boron or mannitol.
* Patients must not have any pre-existing neuropathy of grade > 1.
* Patients must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Female patients who are pregnant or breast feeding or patients of reproductive potential not using an effective method of birth control will be excluded. Women of childbearing potential must have a negative serum pregnancy test within 2 weeks of the first administration of chemo. Also, male patients whose sexual partners are women of child bearing potential not using effective birth control will be excluded.
* Patients with known positivity for human immunodeficiency virus (HIV) will be excluded due to possible pharmacokinetic interactions with bortezomib. Appropriate studies will be undertaken in HIV-positive patients who are receiving or not receiving combination anti-retroviral therapy when indicated.
* Patient must not have received other investigational drugs within 14 days before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios E Argiris, MD, Principal Investigator — Principal Investigator
Locations (21):
- United States (21):
  - UPMC Cancer Center - Teramana Cancer Center - Steubenville, Steubenville, Ohio
  - UPMC Cancer Center - Beaver, Beaver, Pennsylvania
  - UPMC Cancer Center - Clairton, Clairton, Pennsylvania
  - UPMC Cancer Center - Arnold Palmer Pavilion - Greensburg, Greensburg, Pennsylvania
  - UPMC Cancer Center - Oakbrook Commons - Greensburg, Greensburg, Pennsylvania
  - UPMC Cancer Center - Indiana, Indiana, Pennsylvania
  - UPMC Cancer Center - John P. Murtha Pavilion - Johnstown, Johnstown, Pennsylvania
  - UPMC Cancer Center - McKeesport, McKeesport, Pennsylvania
  - UPMC Cancer Center -Haymaker Rd., Monroeville, Pennsylvania
  - UPMC Cancer Center -Mosside Blvd., Monroeville, Pennsylvania
  - UPMC Cancer Center - Sewickley Medical Oncology/Hematology Group, Moon Township, Pennsylvania
  - UPMC Cancer Center -Mt. Pleasant, Mount Pleasant, Pennsylvania
  - UPMC Cancer Center -New Castle, New Castle, Pennsylvania
  - UPMC Cancer Center -Delafield Rd., Pittsburgh, Pennsylvania
  - UPMC Cancer Center - Mercy, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute-Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center - Passavant, Pittsburgh, Pennsylvania
  - UPMC Cancer Center -Drake, Pittsburgh, Pennsylvania
  - UPMC Cancer Center - Uniontown, Uniontown, Pennsylvania
  - UPMC Cancer Center - Washington, Washington, Pennsylvania
  - UPMC Cancer Center -Wexford, Wexford, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib + Doxorubicin: Patients with incurable adenoid cystic carcinoma of the head and neck who received IV bortezomib and doxorubicin
Period: Overall Study
Arm/Group | Bortezomib + Doxorubicin
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib + Doxorubicin
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 56 [44 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is the number participants experiencing partial response (PR) + the number participants experiencing complete response (CR) / the number participants experiencing partial response (PR) + the number participants experiencing complete response (CR) + the number participants experiencing stable disease (SD) + the number participants experiencing progressive disease (PD). RECIST v1.0 criteria for Target Lesions was used: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest s
Time Frame: Up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Bortezomib + Doxorubicin
Number analyzed (Participants) | 9
percentage of participants | 0

2. Primary Outcome: Stable Disease Rate
Description: Using RECIST v1.0 criteria, stable disease rate is the number participants experiencing stable disease (SD) / the number participants experiencing partial response (PR) + the number participants experiencing complete response (CR) + the number participants experiencing stable disease (SD) + the number participants experiencing progressive disease (PD).
Time Frame: Up to 5 years
Population: All patients in this population had stable disease as best response.
Measure: Number; unit: percentage of participants
Arm/Group | Bortezomib + Doxorubicin
Number analyzed (Participants) | 9
percentage of participants | 100

3. Secondary Outcome: Number of Months of Progression-free Survival (PFS)
Description: Number of months that participants experienced stable disease (the disease does not progress per RECIST v1.0 criteria - Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started)
Time Frame: Up to 5 years
Measure: Number; unit: months
Arm/Group | Bortezomib + Doxorubicin
Number analyzed (Participants) | 9
months
  Participant 1 | 8
  Participant 2 | 23
  Participant 3 | 36
  Participant 4 | 4
  Participant 5 | 2
  Participant 6 | 8
  Participant 7 | 26
  Participant 8 | 5
  Participant 9 | 1

4. Secondary Outcome: Number of Months of Survival
Description: Number of months that the participant was alive.
Time Frame: Up to 5 years
Measure: Number; unit: months
Arm/Group | Bortezomib + Doxorubicin
Number analyzed (Participants) | 9
months
  Participant 1 | 29.13
  Participant 2 | 23.40
  Participant 3 | 34.50
  Participant 4 | 8.03
  Participant 5 | 12.20
  Participant 6 | 16.10
  Participant 7 | 25.93
  Participant 8 | 24.97
  Participant 9 | 1.27

5. Secondary Outcome: Median Duration of Stable Disease Response
Description: Median number of months of Stable Disease Response Per RECIST v1.0 (Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started)
Time Frame: Up to 36 months
Measure: Median (Full Range); unit: months
Arm/Group | Bortezomib + Doxorubicin
Number analyzed (Participants) | 9
months | 8 [1 to 36]

ADVERSE EVENTS:
Arm/Group | Bortezomib + Doxorubicin
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib + Doxorubicin (N=9)
Hypotension (Cardiac disorders) | 1
Constipation (General disorders) | 1
Local complication -device/prosthesis-related (Musculoskeletal and connective tissue disorders) | 1
Pain, Abdomen NOS (General disorders) | 1
Pain, Chest/thorax NOS (General disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib + Doxorubicin (N=9)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 5
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 6
Platelets (Blood and lymphatic system disorders) | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2
Sweating (diaphoresis) (General disorders) | 1
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 2
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 3
Hemorrhage, pulmonary/upper respiratory, Nose (Vascular disorders) | 1
Infection - Other (Specify, __) (Infections and infestations) | 2
Opportunistic infection associated with >=Grade 2 Lymphopenia (Infections and infestations) | 1
Edema: limb (Blood and lymphatic system disorders) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 2
Magnesium, serum-low (hypomagnesemia) (Investigations) | 1
Potassium, serum-low (hypokalemia) (Investigations) | 1
Sodium, serum-low (hyponatremia) (Investigations) | 1
Dizziness (Nervous system disorders) | 2
Neuropathy: motor (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 2
Ocular/Visual - Other (Specify, __) (Eye disorders) | 1
Watery eye (epiphora, tearing) (Eye disorders) | 1
Pain - Other (Specify, __) (General disorders) | 1
Pain, Abdomen NOS (General disorders) | 1
Pain, Chest wall (General disorders) | 1
Pain, Extremity-limb (General disorders) | 2
Pain, Head/headache (General disorders) | 3
Pain, Joint (General disorders) | 1
Pain, Pain NOS (General disorders) | 2
Obstruction/stenosis of airway, Bronchus (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1
Urine color change (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No